CLINICAL TRIAL: NCT03934918
Title: Outpatient Cervical Preparation to Reduce Induction Duration in Nulliparous Term Singleton Vertex Women: A Randomized Controlled Trial
Brief Title: Outpatient Cervical Preparation to Reduce Induction Duration in NTSV Women
Acronym: OCPRID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment & funding
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1233410
Record Dates: First submitted 2019-04-18; First posted 2019-05-02 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Cervical Ripening; Outpatient; Patient Satisfaction; Nulliparous; Length of Stay
Keywords: cervical preparation; cervical ripening; NTSV; induction of labor
MeSH Terms: conditions — Patient Satisfaction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Comparing the duration from admission to delivery in nulliparous women between outpatient cervical ripening and those who were admitted for induction of labor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients for IOL with intracervical balloon placed in the outpatient clinic and sent home
  Interventions: Other: Treatment
- Control (No Intervention): Patients for IOL admitted to Labor and Delivery

INTERVENTIONS:
Other: Treatment — Patients for IOL are sent home after placement of intracervical balloon
  Arms: Treatment

SUMMARY:
This study is to compare 2 groups in nulliparous women undergoing cervical ripening for induction of labor. The study hypothesis is that outpatient cervical preparation with a foley catheter can reduce the induction of labor (IOL) time interval from admission to delivery by 50%. A 30 ml transcervical foley catheter is a safe mode of cervical preparation in the outpatient setting, as concluded in Diederen et al, Sciscinoe et al, and Kelly et al. Findings from studies on nulliparous, term, singleton vertex (NTSV) showed patients can be applied to a wide variety of maternity unit sizes as discussed by Main et al. No previous study has evaluated the effectiveness of outpatient cervical preparation in the NTSV population by PUBMED search. Further, no previous study has assessed patient satisfaction cervical preparation in the outpatient setting and no previous study has evaluated whether outpatient cervical preparation has an impact on the length of stay and cost of hospitalization. This study will explore these important questions with the goal of improving current practices in labor induction to be more patient-centered, pragmatic, and cost-effective.

DETAILED DESCRIPTION:
Each participant who is offered an induction of labor from the University of California (UC) Davis Obstetrics and Gynecology clinics will be screened for inclusion criteria. If the participant meets inclusion criteria the participant will be given general information about the study and asked if they would like to participate. If so, research coordinators will meet the participant either during the current clinic visit or a subsequent clinic visit to consent and enroll the participant in the study. During this meeting, the participant will be randomly assigned to Group 1 or Group 2 by using randomization.com and subject number.

Group 1: Treatment

The participant will be given an appointment for fetal monitoring and transcervical foley catheter placement at the Antenatal Testing Unit of the UC Davis Ambulatory Care Center. This may be a same-day appointment. Once the participant presents for her appointment, participant will undergo a routine cervical examination, and routine ultrasound examination for fetal presentation and deep vertical pocket. The participant will also have vitals taken and undergo a brief interview with a provider to rule out rupture of membranes, significant vaginal bleeding, and other perinatal concerns. In order to undergo outpatient cervical preparation, the participant must meet the following criteria: Bishop's score <6 on cervical exam; Normal deep vertical pocket; Cephalic presentation; Negative standard interview to screen for vaginal bleeding, rupture of membranes, labor, and pre-eclampsia; and Blood pressure below 160 bpm systolic and 110 bpm diastolic.

If the participant meets the above criteria for outpatient cervical preparation, a 30 mL transcervical foley catheter will be placed. If the participant does not meet criteria, participant will be sent to Labor and Delivery for possible admission. The participant may elect to receive pain medication intramuscularly for pain management before or after foley catheter placement. After catheter placement the participant will undergo a nonstress test (NST), and if there is no evidence of tachysystole or non-reassuring fetal well-being, participant will be discharged home with a prescription for tylenol. Upon discharge home, the participant will receive instructions on keeping catheter on gentle traction and walking. The participant will be instructed to return once the foley is expelled, or after 24 hours with the foley in place. The participant will also leave with return precautions including rupture of membranes, vaginal bleeding, decreased fetal movement, labor, severe pain, and signs or symptoms of preeclampsia. As a safety measure, the participant will be counseled to call an 24 hour advice nurse line if participant experiences any of the following: Severe pain or discomfort (greater than 8 out of a 10 point scale); Vaginal bleeding; Loss of fluid; Contractions more than 5 minutes apart; Decreased fetal movement; Fevers or chills; Severe headache; Abdominal pain under right rib area; and Spots in vision or blurry vision.

The remaining procedures in this group will follow the standard Labor and Delivery hospital procedures at UC Davis

Group 2: Control The participant will be admitted to Labor and Delivery. The remaining procedures in this group will follow standard Labor and Delivery hospital procedures at UC Davis

The duration anticipated to enroll all study subjects is 10-14 months after Institutional Review Board approval. Approximately 30-40 participant are admitted each month to UC Davis Labor and Delivery. On average, half of these participants are nulliparous. If approximately 5- 10 participants are recruited to each group each month, it will take 10-14 months to reach the goal number of subjects. The duration of an individual subject's participation in the study will be from time of foley catheter insertion (Group 1) or hospital admission time (Group 2) to the time of hospital discharge. Electronic medical records will be accessed during and after this time period only pertaining to the participant's labor including intrapartum and postpartum complications. In addition, participants will be asked survey questions at the time of study enrollment and on postpartum day 1. The estimated date for the investigators to complete this study is two months after enrollment has ended.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women >18 years of age
* Singleton live pregnancy
* Vertex presentation
* Scheduled induction of labor between 37 and 42 weeks gestation
* Bishop score <6

Exclusion Criteria:

* Regular painful contractions (> every 5 minutes)
* Oligohydramnios or anhydramnios
* Breech presentation
* Rupture of membranes
* Fetal heart tracing with minimal variability or significant decelerations with >50% contractions
* Prior vaginal or cesarean delivery
* Contraindication to vaginal delivery (including placenta previa, morbidly adherent placenta, active genital herpes)
* Known or suspected placental abruption
* Major fetal anomaly
* Poorly controlled hypertension (using 2 or more medications; newly diagnosed preeclampsia; preeclampsia with severe features; superimposed preeclampsia)
* Poorly controlled diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Not self described; by virtue of pregnancy
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Duration of time from admission for IOL to delivery | 24 hours
  The time difference from admission to delivery of the infant

SECONDARY OUTCOMES:
Total time of oxytocin use | 24 hours
  time from start to discontinuation prior to delivery
Cesarean delivery | 12 months
  proportion of cesarean section
Blood transfusion | 12 months
  binary - yes or no
Neonatal intensive care unit (NICU) admission | 12 months
  Binary - yes or no
Apgar score at 5 minutes less than 7 | 5 minutes after birth
  Binary - yes or no

OTHER OUTCOMES:
Cost of hospitalization | 12 months
  charges incurred by the patient for all procedures performed including occupancy fees

CONTACTS AND LOCATIONS:
Overall Officials: Herman L Hedriana, MD, Principal Investigator — University of California Davis Health
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Society of Maternal-Fetal (SMFM) Publications Committee. Electronic address: pubs@smfm.org. SMFM Statement on Elective Induction of Labor in Low-Risk Nulliparous Women at Term: the ARRIVE Trial. Am J Obstet Gynecol. 2019 Jul;221(1):B2-B4. doi: 10.1016/j.ajog.2018.08.009. Epub 2018 Aug 9. PMID 30098985
- [Result] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Result] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Result] Kelly AJ, Alfirevic Z, Ghosh A. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2013 Nov 12;(11):CD007372. doi: 10.1002/14651858.CD007372.pub3. PMID 24222365
- [Result] Main EK. Leading Change on Labor and Delivery: Reducing Nulliparous Term Singleton Vertex (NTSV) Cesarean Rates. Jt Comm J Qual Patient Saf. 2017 Feb;43(2):51-52. doi: 10.1016/j.jcjq.2016.11.009. Epub 2016 Nov 15. No abstract available. PMID 28334562
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803